CLINICAL TRIAL: NCT02908594
Title: Institutional Review Board of the Cardinal Tien Hospital
Brief Title: Intradialytic Exercises During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardinal Tien Hospital (Other)
Responsible Party: Principal Investigator, Yueh-Min LIU, Institutional Review Board, Cardinal Tien Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CardinalTH
Record Dates: First submitted 2016-09-10; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Kidney Failure, Chronic
Keywords: Nursing; ESRD; hemodialysis; intradialytic exercise; depression; fatigue; Quality Of Life; self-efficacy; resilience
MeSH Terms: conditions — Kidney Failure, Chronic; Depression; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise group (Experimental): Using the Medical Exercise Peddler 3000, Medi-Bike, Taiwan as an exercise tool. Exercise group received routine care and 3- months exercise. The exercise was performed during the first 2 hr of each haemodialysis session (30 min per session, 3 sessions per week for 3 months).
  Interventions: Device: Medical Exercise Peddler 3000, Medi-Bike, Taiwan
- control group (No Intervention): The control group received routine care

INTERVENTIONS:
Device: Medical Exercise Peddler 3000, Medi-Bike, Taiwan — A horizontal electromagnetic cycle ergometer (Medical Exercise Peddler 3000, Medi-Bike, Taiwan) was used for the exercise program. The cycling equipment includes the resistance of 6 Levels, from Level 1 the lightest to Level 6 the heaviest. Other indicators examined are RPM (rotary per minute), DICT (The distance for this exercise), TIME (The time of exercise). This is the simplest way to use this Motion Exercise Machine. Press the "ST / SP (Start/ Stop)" button to start an exercise program for 30 minutes.
  Arms: exercise group

SUMMARY:
Aim. To investigate the effect of an intradialytic aerobic and resistance cycling exercise program (IARCEP) on depression, fatigue, and quality of life (QOL) in end-stage renal disease (ESRD) patients receiving haemodialysis, and further determine the effect of mediation through self-efficacy and resilience in patients receiving the IARCEP.

Background. Depression and fatigue are common in ESRD patients undergoing haemodialysis, which negatively affects their QOL. Exercise can mitigate this effect. Patient's self-efficacy and resilience may be crucial mediators in exercise.

Design. This study was a randomised controlled trial. Method. Seventy-six participants were randomly assigned to either a control or exercise group. Both groups received routine care; whereas the exercise group participated the 3- months IARCEP. Data were collected at baseline, the first, second, and third months, over a 14 months in 2013-2014.

DETAILED DESCRIPTION:
According to the United States Renal Data System (2015), in 2013, 88.2% of all incident cases of ESRD involved renal replacement therapy with haemodialysis, ESRD is highly prevalent in Taiwan, with 2,902 cases per million people; 89.7% of cases in 2012 involved maintenance haemodialysis treatment as the renal replacement therapy. Patients generally receive haemodialysis 3 days per week, and each session generally takes 4 hr. Beginning dialysis induces multiple physical and psychological stressors in patients. In particular, the importance of intervention programs improving psychosocial function should be noted considering disease and its long-term treatment. High depression and fatigue are crucial for consideration in the global care of dialysis patients because these factors are associated with mortality. A significant correlation exists between reduced physical activity and increased depression or fatigue; with decreased activity, muscle strength decreases, which exacerbates depression and fatigue.

Depression is the most common psychosocial problem observed in ESRD patients undergoing haemodialysis, with a prevalence between 27.9% and 40.2% associated with a high risk of hospitalisation and prolonged hospital stay, reduced quality of life (QOL), decreased adherence to dialysis prescriptions, and increased medical comorbidity.

Fatigue is another critical concern caused by haemodialysis; ESRD patients receiving haemodialysis have reduced red blood cell production, thus causing fatigue, the prevalence of which ranges between 53% and 97%. Fatigue has a negative effect on the physical function, ability to perform daily activities, QOL, and even survival of patients. QOL is the subjective perception of an illness and corresponding treatment regarding physical, psychological, and social well-being; however, QOL serves as a prognostic measure and predictor of survival. ESRD patients receiving haemodialysis have a lower QOL than do other patients with other chronic illnesses and general population. Lower health-related QOL is associated with higher rates of hospitalisation and lower rates of survival among patients undergoing haemodialysis. Therefore, identifying effective interventions to assist ESRD patients receiving haemodialysis in managing their physical, psychological, and social problems is critical.

Regular exercise could improve general health in many chronically ill patients. Planned exercise programs are nonpharmacological interventions that can safely and effectively improve depression, fatigue, and QOL. For ESRD patients undergoing haemodialysis, many previous studies have shown that exercise decreases fatigue and depression, and improves QOL. Accordingly, an intradialytic exercise program should be considered as a possible therapeutic approach for improving fatigue, depression, and QOL in ESRD populations and should be encouraged by and performed in haemodialysis centres. Although the benefits of related exercise programs are known, an effective intradialytic exercise program for routine therapy has not yet been developed. Few previous studies have implemented exercise programs to examine the effects of psychological factors and QOL on patients receiving haemodialysis in Taiwan.

Exercise self-efficacy is a crucial mediator of health behaviour. Self-efficacy is a key construct in social-cognitive theory, in which personal beliefs correspond to an individual's perceived ability to successfully perform specific tasks and activities. Pertaining to beliefs in a person's ability to manage prospective situations, self-efficacy beliefs focus on mediating change in individual behaviours. Thus, self-efficacy has a mediating effect on depression resulting from stressful events. Self-efficacy as a mediator complements family and healthcare provider support in diminishing the negative impact of depression in haemodialysis patients. Relevantly, resilient people tend to have apparent adaptive behaviours, particularly those related to somatic health. Resilience specifically refers to smooth and rapid recovery from setbacks that may occur in a person's life. As such, psychological resilience is considered a protective mechanism that operates in the presence of negative stressors. People who are maladaptive with low competence and low adversity score lower on these measures than resilient and competent groups do. Exercise self-efficacy, resilience, and exercise behaviour are interrelated. Self-efficacy may motivate people to perform their physical activity. However, the true effect of exercise programs fails to account for the mediating effects of exercise self-efficacy and resilience.

Purpose Statements The purpose of this study was to investigate the effect of an intradialytic aerobic and resistance cycling exercise program (IARCEP) on depression, fatigue, and QOL in ESRD patients receiving haemodialysis, and to further determine the effect of mediation through exercise self-efficacy and resilience in patients receiving the IARCEP.

METHODS Research Design and Participants This study adopted a randomised controlled trial design. ESRD participants were recruited from a haemodialysis centre in an 872-bed regional hospital in Northern Taiwan. Data were collected over a 14 months in 2013-2014. The exercise group received routine nursing care in addition to the IARCEP for 3 months. The control group received only routine care in the same study period. A randomisation procedure was performed outside of the study site by two nurse researchers. Permuted-block randomisation, for which every block comprised four patients, was adopted to balance the number of patients in the exercise and control groups. A randomisation list was drawn using random computer-generated sequences. Information regarding these sequences was separately placed in opaque, sealed envelopes to ensure that the participants were randomly allocated to the exercise or control group. Outcomes were repeatedly measured four times at baseline and the first, second, and third months.

Intradialytic aerobic and resistance cycling exercise program (IARCEP) An exercise program brochure for the IARCEP was made available to the exercise group participants to ensure that stationary cycling would be performed appropriately. A horizontal electromagnetic cycle ergometer (Medical Exercise Peddler 3000, Medi-Bike, Taiwan) was used for the participants' cycling performance. The exercise was performed during the first 2 hr of each haemodialysis session (30 min per session, 3 sessions per week for 3 months). All participants were assessed for cardiac and other medical contraindications to exercise by using PAR-Q. Participants were required to perform stationary cycling at an intensity of 11-13 out of 20, corresponding to the rate of perceived exertion on the Borg scale, whereby the intensity was 65%-85% of the participant's maximal capacity, representing the level at which cardiovascular health can be maintained. Exercise was paused when the participants had systolic blood pressure over 180 mmHg, diastolic blood pressure over 95 mmHg, heartbeat under 60 beats/min, or pulse oxyhaemoglobin saturation (SpO2) under 88%. The participants' cardiac rhythm was continuously monitored. Blood pressure and SpO2 was also measured every 5 min. The criteria for interrupting exercise included physical exhaustion, chest pain, dyspnoea, dizziness, and significant instabilities in heartbeat or blood pressure. Immediately following exercise, the participants were assisted with removing the stationary cycling gear to adopt a comfortable position for the immediate assessment of blood pressure, heart rate, and SpO2. Participants were included in the subsequent analysis if they performed the aforementioned exercise procedure at least 10 times per month.

ELIGIBILITY:
Inclusion Criteria:

1. older than 20 years
2. provided consent to participate in this study
3. received haemodialysis 3 times per week for least 3 months
4. missed no more than two dialysis sessions in the previous month
5. had an adequate dialysis, counted by Kt / V over 1.2
6. no lower dialysis graft, basic comprehension and communication in Mandarin or Taiwanese
7. on positive response to any of the supplementary questions in the Physical Activity Readiness Questionnaire (PAR-Q).

Exclusion Criteria:

1. is currently infection or inflammation, autoimmunity disorders, cerebrovascular accidents in the previous 6 months
2. severe muscle weakness or interfering skeletal deformities on lower limbs
3. history of repeated episodes of hypoglycaemia, cardiopulmonary contraindications to resistance exercise (e.g., myocardial infarction, active angina, and uncompensated congestive heart failure in the previous 6 months)
4. lower limb amputation
5. history of participating regularly in exercise programs over 3 months.

Ages: 24 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Generalized estimating equation model on the effects of depression, fatigue, and health-related quality of life | Data were collected over a 14 months in 2013-2014.

SECONDARY OUTCOMES:
Differences-in-differences on the effects of the depression, fatigue, quality of life in exercise group | Data were collected over a 14 months in 2013-2014.
Generalized estimating equation on the mediated effects of self-efficacy and resilience with exercise on outcomes | Data were collected over a 14 months in 2013-2014.
The mediated effects on relationships between exercise and outcomes | Data were collected over a 14 months in 2013-2014.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Ling YEH, Study Director — Professor, Graduate Institute of Integration of Traditional Chinese Medicine with Western Nursing, National Taipei University of Nursing & Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided